CLINICAL TRIAL: NCT02480517
Title: Wave VI Feasibility Study: Phase II Randomized Sham Controlled Study of Renal Denervation for Untreated Stage I and II Hypertension
Brief Title: Sham Controlled Study of Renal Denervation for Untreated Stage I and II Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kona Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KM14-003
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
Keywords: Hypertension; Renal Denervation
MeSH Terms: conditions — Hypertension | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational Therapy (Surround Sound) (Experimental): Investigational Therapy using external focused ultrasound
  Interventions: Device: Ultrasound
- Sham Control (Sham Comparator): Blinded Sham Control Arm
  Interventions: Device: Sham Ultrasound

INTERVENTIONS:
Device: Ultrasound
  Other Names: Surround Sound
  Arms: Investigational Therapy (Surround Sound)
Device: Sham Ultrasound
  Arms: Sham Control

SUMMARY:
The Wave VI study is a, multicenter, prospective, double-blind, randomized, sham controlled feasibility study of the safety of renal denervation in patients with stage I and II hypertension who have an average office systolic blood pressure between 150 and 180 mmHg and have not been on any antihypertensive medications for at least six months.

DETAILED DESCRIPTION:
The primary objective of this feasibility study is to assess the safety of renal denervation using externally focused therapeutic ultrasound with non-invasive targeting for patients with stage I and II hypertension who are not on any antihypertensive medications. The key secondary objective is to assess the effect of the therapy on changes from baseline in ambulatory systolic BP.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age and no more than 80 years of age and can be safely removed from present antihypertensive therapy.
2. Subject has not been taking any anti-hypertensive medications for at least 6 months prior to study enrollment.
3. Subjects must have an average office seated systolic BP (SBP) between 150 mmHg and 180 mmHg inclusive in the untreated state for a minimum of 2 weeks.
4. Mean daytime ambulatory SBP > 135 mmHg and no more than 170 mmHg in addition to mean daytime ambulatory DBP > 85 mmHg.
5. Subject has two functioning kidneys.
6. Subject has an eGFR value of ≥ 30 ml/min/1.73 m² (MDRD formula).

Exclusion Criteria:

a.Any known secondary causes of hypertension.

b.Evidence of current or past history of any clinically significant renal artery stenosis on duplex ultrasound as defined by a finding of at least one of the following:

1. Peak systolic velocity (PSV) in the main renal artery of 150 cm/s or greater;
2. Renal/aortic ratio (RAR) of greater than 3.5; or
3. Complete lack of Doppler signal in any portion of the main renal artery (signifying complete occlusion).

c.Previously documented finding of a 30% or greater renal artery stenosis in any renal arterial vessels as determined by angiographic examination, MRA or CTA.

d.Kidney stones that are 1 cm or greater in size, or that are symptomatic. e.History of intra-abdominal surgery within the past six months or surgery through retroperitoneal path at any time .

f.Previous renal denervation g.Previous renal transplant. h.Heterogeneities in kidney morphology, such as large cysts or tumors (> 2 cm), which are determined at discretion of the investigator to potentially interfere with treatment.

i.Hemodynamically unstable valvular heart disease for which BP reduction would be hazardous in the judgment of the site investigator-physician.

j.Documented history of severe orthostatic hypotension that requires treatment or has necessitated hospitalization.

k.Primary pulmonary hypertension l.History of myocardial infarction, unstable angina pectoris, or cerebrovascular accident within the last six months.

m.BMI over 35 kg/m² and/or mid-arm circumference > 45 cm (creates difficulty with ABPM measurements) n.Anatomy that precludes treatment as determined by the Surround Sound System. This may include any of the following:

1. Target treatment depth as measured by the Surround Sound System of greater than 13 cm (Skin to target);
2. Lack of visualization of the renal artery and or renal artery Doppler signal with the Surround Sound System;
3. Lack of visualization of the renal parenchyma due to obscuration by bowel or other abdominal or retroperitoneal structures; or
4. Narrow window between the superior margin of the iliac crest and the inferior margin of the lowest rib that prevents adequate positioning of both the Surround Sound imaging probe and the treatment unit.

o.Subject is pregnant , nursing, or intends to become pregnant during the study period.

p.Enrollment in another interventional research protocol. q.Any condition that, at the discretion of the investigator, would preclude participation in the study.

r.Subject is unable, or unwilling, to comply with the protocol-required follow-up schedule.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety will be assessed by incidence of Major Adverse Events (MAE), defined as a composite of the following events: | 3 months follow-up
  * All cause mortality;
  * End-stage Renal Disease defined as eGFR < 15 ml/min or need for renal replacement therapy
  * Hospitalization for hypertensive crisis not related to confirmed non-adherence with medications as assessed by toxicological and other medical analyses and testing.
  OR
  - New renal artery stenosis > 70% confirmed by angiography within 3 months of randomization
Change in Office Systolic Blood Pressure (OBP) as measured from screening visit one to the 3 months post randomization follow-up visit. | Baseline and 3 months